CLINICAL TRIAL: NCT00222235
Title: Cognitive and Negative Symptoms in Schizophrenia Trial (CONSIST)
Brief Title: Adjunctive Treatment for Decreasing Symptoms of Schizophrenia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); The Zucker Hillside Hospital (Other); Nathan Kline Institute for Psychiatric Research (Other); University of California, Los Angeles (Other); Sarah Herzog Hospital (Unknown); University of Maryland, College Park (Other)
Responsible Party: Principal Investigator, MPRC, P.I., University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH059807 (NIH); R01MH059807 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; schizoaffective disorder; negative symptoms; cognitive impairments
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Cognitive Dysfunction | interventions — Cycloserine; Glycine

INTERVENTIONS:
Drug: d-cycloserine
Drug: glycine
Drug: placebo

SUMMARY:
This study will determine the effectiveness of treatment with glycine or d-cycloserine in addition to a normal antipsychotic regimen in improving negative symptoms and cognitive impairments in patients with schizophrenia.

DETAILED DESCRIPTION:
A double-blind, placebo controlled clinical trial to examine whether adjunctive treatment with glycine or d-cycloserine, compared to placebo, will improve negative symptoms and cognitive impairments in patients with schizophrenia who remain on their normal antipsychotic regimen.

Multicenter, randomized, double-blinded placebo controlled parallel-groups clinical trial designed to test the hypothesis that interventions (glycine or d-cycloserine) intended to increase glutamatergic activity by action at the NMDA receptor will reduce persistant negative symptoms and cognitive impairments of patients with schizophrenia or schizoaffective disorder. After an initial screening phase to establish clinical stability and eligibility, patients were assigned to one of three adjunctive treatments (placebo, d-cycloserine or glycine)for 16 weeks of double-blind treatment. Patients remained on a stable dose of antipsychotic therapy (other than clozapine) throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of schizophrenia or schizoaffective disorder
* stable, enduring negative symptoms above a certain level (SANS >19)
* clinically stable, with psychotic symptoms measured on BPRS below 19, anxiety/depression on BPRS below 15
* extrapyramidal symptoms measured on SAS below 9
* on stable antipsychotic regimen (not including clozapine)

Exclusion Criteria:

* alcohol or substance dependence within last six months
* alcohol or substance abuse within last month
* organic brain disorder
* medical condition whose pathology or treatment could alter the presentation or treatment of schizophrenia, including active tuberculosis or tuberculosis treatment, kidney stones, and uncontrolled diabetes mellitus
* Female participants could not be pregnant and were required to be using a documented method of contraception.

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240
Dates: Start 2000-01 (Actual); Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
changes from baseline in negative symptoms measured on SANS at 4,8,12 and 16 weeks.
change from baseline on neurocognitive battery measured at 16 weeks.

SECONDARY OUTCOMES:
change in psychotic and depressive symptoms measured at 4,8,12, and 16 weeks.
changes in extrapyramidal side effects at 4,8,12 and 16 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: William T Carpenter, MD, Study Chair — Maryland Psychiatric Research Center, Department of Psychiatry, University of Maryland School of Medicien
Locations (5):
- United States (4):
  - UCLA/VA Greater Los Angeles Health Care System, Los Angeles, California
  - Maryland Psychiatric Research Center, Baltimore, Maryland
  - Zucker Hillside Hospital, Glen Oaks, New York
  - Nathan S Kline Institute for Psychiatric Research, Orangeburg, New York
- Ezrath Nashim Association, Sarah Herzog Memorial Hospital, Jerusalem, Israel

REFERENCES:
- [Derived] Buchanan RW, Javitt DC, Marder SR, Schooler NR, Gold JM, McMahon RP, Heresco-Levy U, Carpenter WT. The Cognitive and Negative Symptoms in Schizophrenia Trial (CONSIST): the efficacy of glutamatergic agents for negative symptoms and cognitive impairments. Am J Psychiatry. 2007 Oct;164(10):1593-602. doi: 10.1176/appi.ajp.2007.06081358. PMID 17898352